CLINICAL TRIAL: NCT04831073
Title: European Registry of Type A Aortic Dissection
Acronym: ERTAAD
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University Hospitals, Leicester (Other); University Hospital Southampton NHS Foundation Trust (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Centre Hospitalier Universitaire de Besancon (Other); Assistance Publique - Hôpitaux de Paris (Other); Ziekenhuis Oost-Limburg (Other); University Hospital Muenster (Other); University of Hamburg-Eppendorf (Other); Institute for Clinical and Experimental Medicine (Other Government); Northern General Hospital, Herries Road, Sheffield (Unknown); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); University Hospital, Udine, Italy (Other); Heart Center Leipzig - University Hospital (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); AZ Sint-Jan AV (Other); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); University of Turin, Italy (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Fausto Biancari, Professor, Helsinki University Central Hospital
Other Study IDs: 100968
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Type A Aortic Dissection
Keywords: Aortic dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute type A aortic dissection: Patients who underwent surgery for acute type A aortic dissection
  Interventions: Procedure: Surgery on the ascending aorta with or without repair of the aortic root and/or aortic arch

INTERVENTIONS:
Procedure: Surgery on the ascending aorta with or without repair of the aortic root and/or aortic arch — Surgical repair of the ascending aorta with or without surgical repair of the aortic root and/or aortic arch

SUMMARY:
Acute Stanford type A aortic dissection (TAAD) is a life-threatening condition. Surgery is usually performed as a salvage procedure and is associated with significant postoperative early mortality and morbidity. Understanding the patient's conditions and treatment strategies which are associated with these adverse events is essential for an appropriate management of acute TAAD.

DETAILED DESCRIPTION:
Twenty centers from eight European centers of cardiac surgery have collaborated to create a multicentre observational registry (ERTAAD), which will enroll consecutive patients who underwent surgery for acute TAAD from January 2005 to March 2021. The investigators will compare patient's comorbidities, condition at referral, surgical strategies and perioperative treatments in patients with and without early and late adverse events. The primary clinical outcome will be in-hospital mortality, late mortality and reoperations on the aorta. Secondary outcomes will be stroke, acute kidney injury, surgical site infection, reoperation for bleeding, transfusion of blood products and length of stay in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Type A aortic dissection or intramural hematoma involving the aortic root/ascending aorta;
* Patients aged > 18 years:
* Symptoms started within 7 days from surgery;
* Primary surgical repair of acute type A aortic dissection;
* Any other major cardiac surgical procedure concomitant with surgery for type A aortic dissection.

Exclusion Criteria:

* Patients aged < 18 years;
* Onset of symptoms > 7 days from surgery;
* Prior procedure for type A aortic dissection;
* Retrograde type A aortic dissection (with primary tear located in the descending aorta);
* Concomitant endocarditis;
* Type A aortic dissection secondary to blunt or penetrating chest trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical repair for acute type A aortic dissection or intramural hematoma involving the aortic root/ascending aorta.
Sampling Method: Non-Probability Sample
Enrollment: 3902 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Mortality rate | During the index hospital stay until last follow-up control
  All-cause mortality
Cumulative incidence of reoperation on the aorta | During the index hospital stay until last follow-up control
  Any surgical and endovascular procedure on any segment of the aorta for aortic dissection or its related complication

SECONDARY OUTCOMES:
Incidence of stroke | From date of procedure until the date of hospital discharge, assessed up to 3 months
  change in the level of consciousness, hemiplegia, hemiparesis, numbness, or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopia, amaurosis fugax, or other neurological signs or symptoms consistent with stroke duration of a focal or global neurological deficit ≥ 24 h; OR <24 h if available neuroimaging documents a new brain hemorrhage or infarct; OR the neurological deficit results in death.
Incidence of acute kidney injury | From date of procedure until the date of hospital discharge, assessed up to 3 months
  It will be defined according to postoperative change in serum creatinine levels and its severity will be stratified according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Incidence of surgical site infection | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Proven infection involving deep sternal wound tissues and/or mediastinum.
Incidence of reoperation for bleeding | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Chest reopening for excessive bleeding.
Incidence and amount of blood transfusion | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Transfusions of red blood cells
Length of stay in the intensive care unit | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Duration of stay in the intensive care unit
Incidence of global brain ischemia | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Diffuse hypoxic damage as diagnosed at brain imaging and electroencephalography.
Incidence of paraplegia/paraparesis | From date of procedure until the date of hospital discharge, assessed up to 3 months
  Bilateral weakness and/or multimodality sensory disturbance below the level of the ischemic spinal lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Biancari, Principal Investigator — Helsinki University Hospital, Helsinki, Finland
Locations (20):
- Belgium (5):
  - AZ St-Jan, Bruges
  - Saint-Luc's Hospital, Brussels
  - University Hospital Antwerp, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospitals Leuven, Leuven
- Institute of Clinical and Experimental Medicine, Prague, Czechia
- Helsinki University Hospital, Helsinki, Finland
- France (2):
  - Henri Mondor University Hospital, Créteil, Paris
  - University Hospital Jean Minjoz, Besançon
- Germany (3):
  - University Heart & Vascular Centre Hamburg, Hamburg
  - Leipzig Heart Center, Leipzig
  - Münster University Hospital, Münster
- Italy (3):
  - University of Torino, Torino
  - University of Udine, Udine
  - University of Verona Medical School, Verona
- Hospital Clínic de Barcelona, Barcelona, Spain
- United Kingdom (4):
  - University Hospitals of Leicester, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Northern General Hospital, Sheffield
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demal TJ, Knochenhauer T, Weimann J, Juvonen T, Makikallio T, Fiore A, Perrotti A, Pettinari M, Peterss S, Buech J, Radner C, Dell'Aquila AM, Wisniewski K, Pol M, Kacer P, Onorati F, Francica A, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Lega JR, Pinto AG, Acharya M, Field M, Kuduvalli M, Nappi F, Gerelli S, Di Perna D, Gatti G, Mazzaro E, Rosato S, D'Errigo P, Mariscalco G, El-Dean Z, Detter C, Reichenspurner H, Polvani G, Biancari F, Conradi L. Outcome after day- and nighttime surgery for acute type A aortic dissection. Eur J Cardiothorac Surg. 2025 Jun 3;67(6):ezaf192. doi: 10.1093/ejcts/ezaf192. PMID 40569847
- [Derived] Biancari F, Makikallio T, Rosato S, Juvonen T, Mariscalco G, El-Dean Z, Acharya M, Pettinari M, Rodriguez-Lega J, Pinto AG, Perrotti A, Onorati F, Wisniewski K, Conradi L, Demal T, Pol M, Rocek J, Kacer P, Gatti G, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Peterss S, Buech J, Radner C, Field M, Harky A, Fiore A, Senemaud J, Mustonen C, Dell'Aquila AM, D'Errigo P, Polvani G, Di Perna D. Carotid artery dissection and neurological complications after surgery for type 1 aortic dissection. Open Heart. 2025 Mar 12;12(1):e002882. doi: 10.1136/openhrt-2024-002882. PMID 40081929
- [Derived] Biancari F, Fileccia D, Ferrante L, Makikallio T, Juvonen T, Jormalainen M, Mariscalco G, El-Dean Z, Pettinari M, Rodriguez Lega J, Pinto AG, Perrotti A, Onorati F, Wisniewski K, Demal T, Kacer P, Rocek J, Di Perna D, Vendramin I, Piani D, Rinaldi M, Quintana E, Pruna-Guillen R, Peterss S, Buech J, Radner C, Kuduvalli M, Harky A, Fiore A, D'Alonzo M, Dell'Aquila AM, Gatti G, Conradi L, Ballotta A, Field M. Extent of surgical repair and outcomes after surgery for type A aortic dissection. BJS Open. 2025 Mar 4;9(2):zraf003. doi: 10.1093/bjsopen/zraf003. PMID 40071739
- [Derived] Biancari F, Gatti G, Makikallio T, Juvonen T, Mariscalco G, El-Dean Z, Pettinari M, Rodriguez Lega J, Perrotti A, Onorati F, Wisniewki K, Demal T, Kacer P, Perna DD, Vendramin I, Rinaldi M, Ferrante L, Quintana E, Buech J, Radner C, Fiore A, Dell'Aquila AM, D'Errigo P, Rosato S, Polvani G, Peterss S. Ascending aortic replacement versus aortic root replacement in patients with type A aortic dissection involving the aortic root. Ther Adv Cardiovasc Dis. 2025 Jan-Dec;19:17539447241303408. doi: 10.1177/17539447241303408. PMID 39840731
- [Derived] Biancari F, Lega JR, Mariscalco G, Peterss S, Buech J, Fiore A, Perrotti A, Rukosujew A, Pinto AG, Demal T, Wisniewski K, Pol M, Gatti G, Vendramin I, Rinaldi M, Pruna-Guillen R, Di Perna D, El-Dean Z, Sherzad H, Nappi F, Field M, Pettinari M, Jormalainen M, Dell'Aquila AM, Onorati F, Quintana E, Juvonen T, Makikallio T. Aortic arch surgery for DeBakey type 1 aortic dissection in patients aged 60 years or younger. BJS Open. 2024 May 8;8(3):zrae047. doi: 10.1093/bjsopen/zrae047. PMID 38768283
- [Derived] Juvonen T, Vendramin I, Mariscalco G, Jormalainen M, Perrotti A, Herve A, Mazzaro E, Gatti G, Pettinari M, Peterss S, Buech J, Nappi F, Pinto AG, Rodriguez Lega J, Pol M, Rocek J, Kacer P, Rukosujew A, Wisniewski K, Piani D, Demal T, Conradi L, Ferrante L, Rinaldi M, Quintana E, Pruna-Guillen R, Gerelli S, Di Perna D, Fiore A, Folliguet T, Acharya M, El-Dean Z, Field M, Kuduvalli M, Onorati F, Francica A, Makikallio T, Dell'Aquila AM, Mustonen C, Raivio P, Rosato S, Biancari F. Femoral arterial cannulation for surgical repair of stanford type A aortic dissection. World J Surg. 2024 Jul;48(7):1771-1782. doi: 10.1002/wjs.12203. Epub 2024 Apr 30. PMID 38686961
- [Derived] Biancari F, Onorati F, Peterss S, Buech J, Mariscalco G, Lega JR, Pinto AG, Fiore A, Perrotti A, Herve A, Rukosujew A, Demal T, Conradi L, Wisniewski K, Pol M, Kacer P, Gatti G, Mazzaro E, Vendramin I, Piani D, Rinaldi M, Ferrante L, Pruna-Guillen R, Di Perna D, Gerelli S, El-Dean Z, Nappi F, Field M, Kuduvalli M, Pettinari M, Francica A, Jormalainen M, Dell'Aquila AM, Makikallio T, Juvonen T, Quintana E. Nature of Neurological Complications and Outcome After Surgery for Type A Aortic Dissection. Am J Cardiol. 2024 May 15;219:85-91. doi: 10.1016/j.amjcard.2024.03.001. Epub 2024 Mar 6. PMID 38458584
- [Derived] Biancari F, Perrotti A, Juvonen T, Mariscalco G, Pettinari M, Lega JR, Di Perna D, Makikallio T, Onorati F, Wisniewki K, Demal T, Pol M, Gatti G, Vendramin I, Rinaldi M, Quintana E, Peterss S, Field M, Fiore A. Diameter and dissection of the abdominal aorta and the risk of distal aortic reoperation after surgery for type A aortic dissection. Int J Cardiol. 2024 Jun 1;404:131938. doi: 10.1016/j.ijcard.2024.131938. Epub 2024 Mar 7. PMID 38458387
- [Derived] Biancari F, Demal T, Nappi F, Onorati F, Francica A, Peterss S, Buech J, Fiore A, Folliguet T, Perrotti A, Herve A, Conradi L, Rukosujew A, Pinto AG, Lega JR, Pol M, Rocek J, Kacer P, Wisniewski K, Mazzaro E, Vendramin I, Piani D, Ferrante L, Rinaldi M, Quintana E, Pruna-Guillen R, Gerelli S, Di Perna D, Acharya M, Mariscalco G, Field M, Kuduvalli M, Pettinari M, Rosato S, D'Errigo P, Jormalainen M, Mustonen C, Makikallio T, Dell'Aquila AM, Juvonen T, Gatti G. Baseline risk factors of in-hospital mortality after surgery for acute type A aortic dissection: an ERTAAD study. Front Cardiovasc Med. 2024 Jan 15;10:1307935. doi: 10.3389/fcvm.2023.1307935. eCollection 2023. PMID 38288052
- [Derived] Juvonen T, Jormalainen M, Mustonen C, Demal T, Fiore A, Perrotti A, Herve A, Mazzaro E, Gatti G, Pettinari M, Peterss S, Buech J, Nappi F, Conradi L, Pinto AG, Rodriguez Lega J, Pol M, Kacer P, Dell'Aquila AM, Rukosujew A, Wisniewski K, Vendramin I, Piani D, Ferrante L, Rinaldi M, Quintana E, Pruna-Guillen R, Gerelli S, Di Perna D, Folliguet T, Acharya M, Field M, Kuduvalli M, Onorati F, Rossetti C, Makikallio T, Raivio P, Mariscalco G, Biancari F. Direct Aortic Versus Supra-Aortic Arterial Cannulation During Surgery for Acute Type A Aortic Dissection. World J Surg. 2023 Nov;47(11):2899-2908. doi: 10.1007/s00268-023-07116-z. Epub 2023 Jul 11. PMID 37432422
- [Derived] Biancari F, Juvonen T, Fiore A, Perrotti A, Herve A, Touma J, Pettinari M, Peterss S, Buech J, Dell'Aquila AM, Wisniewski K, Rukosujew A, Demal T, Conradi L, Pol M, Kacer P, Onorati F, Rossetti C, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Rodriguez Lega J, Pinto AG, Acharya M, El-Dean Z, Field M, Harky A, Nappi F, Gerelli S, Di Perna D, Gatti G, Mazzaro E, Rosato S, Raivio P, Jormalainen M, Mariscalco G. Current Outcome after Surgery for Type A Aortic Dissection. Ann Surg. 2023 Oct 1;278(4):e885-e892. doi: 10.1097/SLA.0000000000005840. Epub 2023 Mar 13. PMID 36912033
- [Derived] Biancari F, Dell'Aquila AM, Gatti G, Perrotti A, Herve A, Touma J, Pettinari M, Peterss S, Buech J, Wisniewski K, Juvonen T, Jormalainen M, Mustonen C, Rukosujew A, Demal T, Conradi L, Pol M, Kacer P, Onorati F, Rossetti C, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Lega JR, Pinto AG, Acharya M, El-Dean Z, Field M, Harky A, Kuduvalli M, Nappi F, Gerelli S, Di Perna D, Mazzaro E, Rosato S, Fiore A, Mariscalco G. Interinstitutional analysis of the outcome after surgery for type A aortic dissection. Eur J Trauma Emerg Surg. 2023 Aug;49(4):1791-1801. doi: 10.1007/s00068-023-02248-2. Epub 2023 Feb 24. PMID 36826589
- [Derived] Biancari F, Mariscalco G, Yusuff H, Tsang G, Luthra S, Onorati F, Francica A, Rossetti C, Perrotti A, Chocron S, Fiore A, Folliguet T, Pettinari M, Dell'Aquila AM, Demal T, Conradi L, Detter C, Pol M, Ivak P, Schlosser F, Forlani S, Chetty G, Harky A, Kuduvalli M, Field M, Vendramin I, Livi U, Rinaldi M, Ferrante L, Etz C, Noack T, Mastrobuoni S, De Kerchove L, Jormalainen M, Laga S, Meuris B, Schepens M, El Dean Z, Vento A, Raivio P, Borger M, Juvonen T. European registry of type A aortic dissection (ERTAAD) - rationale, design and definition criteria. J Cardiothorac Surg. 2021 Jun 10;16(1):171. doi: 10.1186/s13019-021-01536-5. PMID 34112230